CLINICAL TRIAL: NCT01967485
Title: Text Messaging Adherence to Stimulant Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Mai Uchida, Child Psychiatrist, Pediatric Psychopharmacology and Adult ADHD Program, Massachusetts General Hospital; Instructor in Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-P-002161
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Medication adherence; Disease management; Text message; ADHD; Children; Reminder systems; Text Messaging; Telemedicine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Medication Adherence | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Messaging (Experimental): Text messaging to the parents of children. Children will receive open treatment for Attention Deficit/Hyperactivity Disorder (ADHD) with stimulant medication.
  Interventions: Other: Text- Messaging; Other: Treatment as usual
- No Text Messaging (Active Comparator): Children will receive open treatment for ADHD with stimulant medication. This group will not get the text messaging intervention, but will receive treatment as usual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Text- Messaging — Text messages will be sent to the parents of children enrolled in the study.
  Arms: Text Messaging
Other: Treatment as usual — Children will receive stimulant treatment for ADHD.

SUMMARY:
The purpose of this study is to determine if an individualized text messaging intervention for the parents of children with Attention Deficit/Hyperactivity Disorder is effective in improving medication adherence and disease management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ages 6-17 years
* A diagnosis of ADHD (inattentive, hyperactive/impulsive, or combined type) according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) based on clinical assessment and supported by a Clinical Global Impression- ADHD (CGI-ADHD) Severity Score of at least 4 (Moderately Ill)
* Has a parent in possession of a cellular phone with text messaging capabilities and is interested in and willing to receive planned text messages
* Has never been treated with stimulant medication, or has begun treatment with stimulant medication within three months of study enrollment.

Exclusion Criteria:

* Any serious, unstable, chronic medical condition, per clinician assessment
* Cardiovascular disease
* Current or past history of seizures
* Treatment with stimulant medication beyond three months prior to enrollment
* Pregnant or nursing females
* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild
* Unstable psychiatric illness other than ADHD, including, but not limited to: Autism, Bipolar Disorder, Psychosis, Major Depressive Disorder, Anorexia, Bulimia, Post-Traumatic Stress Disorder and Anxiety Disorders
* History of multiple adverse drug reactions
* Presence of suicidal risk, or homicidality
* Unwilling/unable to comply with study procedures
* Poor command of the English language

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | Six Months
  Adherence to the individualized medication regimen

CONTACTS AND LOCATIONS:
Overall Officials: Mai Uchida, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No